CLINICAL TRIAL: NCT07130513
Title: The Effect of Krill Oil Supplementation on Muscle Function in Adults With High-risk Long-term Conditions: a Randomized Controlled Pilot Study.
Brief Title: Investigating the Feasibility of Krill Oil Intervention to Improve Muscle Function in Adults With Long-term Conditions
Acronym: KOMM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Stuart Gray, Professor Stuart Gray, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KOMM
Record Dates: First submitted 2025-08-04; First posted 2025-08-19 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Krill Oil; Muscle Function; Grip Strength; Long-Term Conditions; Omega 3 Fatty Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Krill Oil group (Experimental): 4 g/day of krill oil (Superba™ Antarctic Krill Oil, 1000 mg capsules) for 12 weeks.
  Interventions: Dietary Supplement: Krill oil supplementation
- Arm 2: Control group (Placebo Comparator): 4 g/day of placebo (vegetable oil capsules) for 12 weeks.
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Krill oil supplementation — Krill oil supplementation program providing 4 g/day of krill oil (Superba™ Antarctic Krill Oil, 1000 mg capsules) for 12 weeks.
  Other Names: Omega 3 supplementation
  Arms: Arm 1: Krill Oil group
Dietary Supplement: Control — Vegetable oil supplementation (4 g/day)
  Arms: Arm 2: Control group

SUMMARY:
This study will recruit 30 adults (men and women, aged 18 years and over) who will be randomly assigned to one of two groups in a 12-week double-blind pilot trial. Participants will receive either:

* Arm 1: Krill Oil group: 4 g/day of krill oil supplements (Superba™ Antarctic Krill Oil, 1000 mg capsules), or
* Arm 2: Control group: 4 g/day of placebo (vegetable oil capsules).

Participants will be instructed to maintain their usual diet and physical activity patterns throughout the study.

Eligibility will be assessed using a health screening questionnaire, completed with the researcher's assistance, before obtaining informed consent. Habitual physical activity will be evaluated using the International Physical Activity Questionnaire (short form), and dietary intake will be assessed with the EPIC Food Frequency Questionnaire (FFQ) at both the beginning and end of the study. In addition, participants will record their fish consumption weekly using a dedicated logbook.

Measurements will be taken at baseline and after 12 weeks, including:

* Blood samples to assess inflammatory and metabolic markers.
* Anthropometry and body composition, including weight, height, fat mass, fat percentage, and muscle mass (via ultrasound).
* Muscle strength, measured using handgrip strength and maximal voluntary contraction (each performed three times with rest between attempts).
* Physical performance, assessed with a 4-meter walk test at normal speed Upon completing the study, participants will receive a £50 voucher in appreciation of their contribution.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥18 years who are in the high-risk long-term condition group (having one or more LTCs, including rheumatoid arthritis, gout, type 2 diabetes, coronary heart disease, and stroke [including transient ischemic attack, TIA]).

Exclusion Criteria:

* Participants are diagnosed with and being treated for any type of cancer.
* Presence of neurocognitive disorders or any health condition affecting memory (e.g., Alzheimer's disease, dementia).
* Aortic stenosis, history of haemorrhagic stroke, or presence of aneurysms.
* Current anticoagulant therapy.
* Use of any muscle mass supplements or presence of physiological conditions such as pregnancy or breastfeeding.
* History of allergy to fish or fish oil.
* Regular consumption of more than one portion of oily fish per week, or use of fish oil or krill oil supplements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Grip strength | Changes from baseline to week 12
  Measured using a handgrip dynamometer

SECONDARY OUTCOMES:
Knee extendor Strength | Changes from baseline to week 12
  Knee extensor maximal torque measured during an isometric maximal voluntary contraction (MVC)
Muscle size, assessed as vastus lateralis muscle thickness by ultrasound | Changes from baseline to week 12
  The investigators will assess vastus lateralis muscle thickness using B-mode ultrasound, with participants in a supine position. This measurement will also serve as an indirect indicator of muscle damage through cell swelling. The measurement site will be located at 10% of the thigh circumference lateral to the midpoint between the iliac crest and the superior border of the patella.
Gait speed | From baseline to week 12
  Gait speed will be assessed as a measure of physical function.
Fatty Acid Composition | From baseline to week 12
  A venous blood sample (15 ml) will be collected from an antecubital vein by a trained member of the research team and analysed for erythrocyte fatty acid profile.
Inflammatory and metabolic markers | From baseline to week 12
  A venous blood sample (15 ml) will be collected by a trained member of the research team from an antecubital vein and analysed to estimate plasma glucose, lipids (triacylglycerol, total cholesterol, HDL), and markers of inflammation (e.g., hsCRP, IL-6, TNF-α, homocysteine).
Height | Changes from baseline to week 12
  Height recorded using a stadiometer in centimetre at the beginning of the study.
Bodyweight | Changes from baseline to week 12
  Changes in bodyweight, recorded in kilogram. Measured via body composition analyser.
Body Mass Index (BMI) | Changes from baseline to week 12
  Will be calculated from the bodyweight (in kilogram) and height (in meter) according to the BMI formula (kg/m^2).
Body Fat Mass | Changes from baseline to week 12
  Changes in body fat mass, recorded in kilogram. Measured via body composition analyser.
Body Fat Percentages | Changes from baseline to week 12
  Changes in body fat percentage, recorded in percentage. Measured via body composition analyser.
Fat Free Mass | Changes from baseline to week 12
  Changes in fat free mass, recorded in kilogram. Measured via body composition analyser.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Lab 242, Sir James Black Building, University of Glasgow, Glasgow, Lanarkshire
  - University of Glasgow, Glasgow, Lanarkshire

IPD SHARING:
Plan to Share IPD: No